CLINICAL TRIAL: NCT00628810
Title: Chemotherapy With FOLFIRI Plus Bevacizumab (AvastinR) in Patients With Metastatic Colorectal Cancer Bearing Genotype UGT1A1*1/UGT1A1*1 or UGT1A1*1/UGT1A1*1/UGT1A1*28: Prospective, Phase II, Multicenter Study
Brief Title: Combination Chemotherapy and Bevacizumab in Treating Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000564065; FFCD-0504; EUDRACT-2006-003157-25; EU-20755
Record Dates: First submitted 2008-03-04; First posted 2008-03-05 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; adenocarcinoma of the rectum; stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Bevacizumab; Fluorouracil; Irinotecan; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI fort plus bevacizumab (Experimental): Bevacizumab 5 mg/kg D1, irinotecan 260 mg/m2 D1, LV 400 mg/m2 D1, 5FU 400 mg/m2 IV bolus D1, and 5FU 2,400 mg/m2 46-hour infusion D1-2 every 2 weeks. Treatment was started within 2 weeks after inclusion in the study.
  Interventions: Biological: bevacizumab; Drug: fluorouracil; Drug: irinotecan hydrochloride; Drug: leucovorin calcium

INTERVENTIONS:
Biological: bevacizumab
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving combination chemotherapy together with bevacizumab may kill more tumor cells.

PURPOSE: This phase II trial is studying the side effects of giving combination chemotherapy together with bevacizumab and to see how well it works in treating patients with metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the objective response (RECIST criteria) at 6 months associated with FOLFIRI and bevacizumab therapy.
* Evaluate the tolerability (NCI CTC v. 2.0 criteria) of this treatment.

Secondary

* Evaluate progression-free survival and overall survival.
* Determine the time to treatment failure.
* Evaluate the quality of life (EuroQOL EQ5D questionnaire).
* Explore the prognostic factors associated with the tolerability and efficacy of this treatment.

OUTLINE: This is a multicenter study. Patients are stratified according to genotype (UCT1A1*1/ UCT1A1*1 vs UCT1A1*1/ UCT1A1*28).

Patients receive bevacizumab IV over 30-90 minutes, irinotecan hydrochloride IV over 90 minutes, leucovorin calcium IV over 2 hours, and fluorouracil IV over 46 hours on day 1. Treatment repeats every 2 weeks in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, every 4 courses, and then every 2 months after the completion of study therapy.

After completion of study therapy, patients are followed every 2-3 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of metastatic adenocarcinoma of the colon or rectum

  * Not curable by surgery
* Genotype UGT1A1*1/UGT1A1*1 or UGT1A1*1/ UGT1A1*28
* Measurable disease
* No original tumor in place
* No secondary cerebral metastases

PATIENT CHARACTERISTICS:

Inclusion criteria:

* WHO performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm3
* Platelet count ≥ 100,000/mm3
* Hemoglobin ≥ 9.0 g/dL
* Total bilirubin ≤ 1.5 times normal
* Alkaline phosphatase ≤ 2.5 times normal (5 times normal if liver involvement)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients of must use effective contraception

Exclusion criteria:

* Progressive gastrointestinal ulcer, hemorrhagic ulcer, or perforation in the past 6 months
* Enteropathy or chronic diarrhea
* Proteinuria > 500 mg/24 hours
* Active cardiac disease
* Uncontrolled hypertension
* Myocardial infarction in the past 12 months
* Angina
* NYHA grade II-IV congestive heart disease
* Severe arrhythmia even with treatment
* Peripheral vascular disease ≥ grade II
* Nonhealing wound, ulcer, or severe bone fracture
* Hemorrhagic diatheses or coagulopathy
* Severe or uncontrolled infection
* Severe or uncontrolled medical condition
* Other malignant disease in the past 5 years except curatively treated basal cell skin cancer or carcinoma in situ of the uterine cervix
* Severe traumatic injury within the past 4 weeks

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy for metastatic disease

  * One prior regimen of chemotherapy in the neoadjuvant or adjuvant setting for the original tumor allowed
* At least 6 months since prior chemotherapy
* No prior irinotecan hydrochloride or bevacizumab
* No oral or parenteral anticoagulant therapy within the past 10 days

  * Warfarin allowed provided INR < 1.5
* No major surgery or biopsy within the past 4 weeks
* No puncture in the past 7 days
* No planned major surgery
* No concurrent daily or chronic aspirin (> 325 mg/day), anti-inflammatories, or steroids
* No other concurrent anticancer therapy

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Objective response at 6 months by RECIST | 6 months
Tolerability evaluated by NCI CTC v. 2.0 criteria | From Inclusion

SECONDARY OUTCOMES:
Progression-free and overall survival | From Inclusion
Time to treatment failure | From Inclusion
Quality of life using the EuroQOL EQ5D questionnaire | From Inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Martina Schneider, Study Chair — Federation Francophone de Cancerologie Digestive
Locations (32):
- France (32):
  - Centre Hospitalier d'Abbeville, Abbeville
  - Centre Hospitalier Universitaire d'Amiens, Amiens
  - Hopital Duffaut, Avignon
  - C.H.G. Beauvais, Beauvais
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hopital Ambroise Pare, Boulogne-Billancourt
  - Centre Hospitalier Pierre Oudot, Bourgoin
  - Centre Hospitalier General, Brivé
  - CHU de Caen, Caen
  - Centre Regional Francois Baclesse, Caen
  - Centre Hospitalier de Chalons-en-Champagne, Châlons-en-Champagne
  - Hopitaux Civils de Colmar, Colmar
  - Hopital Du Bocage, Dijon
  - Federation Francophone de Cancerologie Digestive, Dijon
  - Clinique Saint Vincent, Épernay
  - Centre Hospitalier Departemental, La Roche-sur-Yon
  - Hopital Andre Mignot, Le Chesnay
  - Centre Hospitalier Universitaire de Bicetre, Le Kremlin-Bicêtre
  - CHU de la Timone, Marseille
  - CHU Nord, Marseille
  - Hopital de l'Archet CHU de Nice, Nice
  - CHR D'Orleans - Hopital de la Source, Orléans
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat - Claude Bernard, Paris
  - CHU - Robert Debre, Reims
  - Hopital Charles Nicolle, Rouen
  - Clinique Mathilde, Rouen
  - Clinique Armoricaine De Radiologie, Saint-Brieuc
  - CHRU de Tours - Hopital Trousseau, Tours
  - Centre Hospitalier General Lucien Hussel, Vienne
  - Clinique du Tonkin, Villeurbanne

REFERENCES:
- [Result] Manfredi S, Bouche O, Rougier P, Dahan L, Loriot MA, Aparicio T, Etienne PL, Lafargue JP, Lecaille C, Legoux JL, Le Malicot K, Maillard E, Lecomte T, Khemissa F, Breysacher G, Michel P, Mitry E, Bedenne L. High-Dose FOLFIRI plus Bevacizumab in the Treatment of Metastatic Colorectal Cancer Patients with Two Different UGT1A1 Genotypes: FFCD 0504 Study. Mol Cancer Ther. 2015 Dec;14(12):2782-8. doi: 10.1158/1535-7163.MCT-15-0293. Epub 2015 Oct 22. PMID 26494856